CLINICAL TRIAL: NCT04638088
Title: Comparison of Radical Prostatectomy for the Treatment of Prostate Cancer, Performed by Robot-assisted or Standard Laparoscopy or by Laparotomy : a Multicentric Prospective Study.
Brief Title: Comparison of Radical Prostatectomy Performed by Robot-assisted Laparoscopy or Conventional Laparoscopy or by Laparotomy
Acronym: EMUPRO
Status: Recruiting | Type: Observational
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Other Study IDs: GCS-ELSAN-0620
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Prostate Cancer
Keywords: robot-assisted laparoscopy; laparotomy; conventional laparoscopy; prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- robot-assisted laparoscopy: radical prostatectomy performed by robot-assisted laparoscopy
  Interventions: Other: assessment of urinary function and erectil function before and after prostatectomy
- conventional laparoscopy: radical prostatectomy performed by conventional laparoscopy
  Interventions: Other: assessment of urinary function and erectil function before and after prostatectomy
- laparotomy: radical prostatectomy performed by laparotomy
  Interventions: Other: assessment of urinary function and erectil function before and after prostatectomy

INTERVENTIONS:
Other: assessment of urinary function and erectil function before and after prostatectomy — assessment of urinary function and erectil function before and after prostatectomy performed by robot assisted or conventional laparoscopy or laparotomy will complete

SUMMARY:
Minimally invasive surgery has developed widely since the 1980s and has revolutionized the practices of surgeons. In urology, the development of laparoscopy and then robot-assisted surgery has considerably improved the management of pathologies. In France, as in all the countries concerned, the spread of robotic surgery has taken place without prior studies validating this new technology, nor organizational rules in terms of quality and access to care. The report of the Haute Autorité de Santé dated November 2016 underlines the weakness of the methodological quality of studies and meta-analyzes evaluating robot-assisted total prostatectomy compared to other surgical techniques by laparotomy or conventional laparoscopy. It therefore appears important to evaluate in a large study the interest of this technique in order to help the authorities to decide on the real benefit of this technology and to provide reliable answers to the patients.

DETAILED DESCRIPTION:
Minimally invasive surgery has developed widely since the 1980s and has revolutionized the practices of surgeons. In urology, the development of laparoscopy and then robot-assisted surgery has considerably improved the management of pathologies. In France, as in all the countries concerned, the spread of robotic surgery has taken place without prior studies validating this new technology, nor organizational rules in terms of quality and access to care. The report of the Haute Autorité de Santé dated November 2016 underlines the weakness of the methodological quality of studies and meta-analyzes evaluating robot-assisted total prostatectomy compared to other surgical techniques by laparotomy or conventional laparoscopy. It therefore appears important to evaluate in a large study the interest of this technique in order to help the authorities to decide on the real benefit of this technology and to provide reliable answers to the patients.

ELIGIBILITY:
Inclusion Criteria:

* patient hospitalized for a planned radical prostatectomy

Exclusion Criteria:

* Consent refusal from the patient
* Patients protected by law (Art.L 1121-5, 1121-6, 1121-8 du Code de la santé publique)
* Absence of a French Health Care Insurance coverage

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient hospitalized for a planned radical prostactectomy .
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2025-04-22 (Estimated); Study Completion 2030-04-22 (Estimated)

PRIMARY OUTCOMES:
Impact of the prostatectomy procedure (robot assisted laparoscopy, conventional laparoscopy and surgical laparotomy) on the urinary function assessed by the EPIC 50 score | 45 Days after the surgery
  Comparison of the prostatectomy performed by robot assisted laparoscopy or conventional laparoscopy and by surgical laparotomy on the urinary function assessed by the EPIC 50 score (Expanded Prostate Cancer Index Composite)

SECONDARY OUTCOMES:
impact of the robot assisted laparoscopy compared to conventional laparoscopy and by surgical laparotomy in radical prostatectomy on the erectile function assessed by the EPIC 50 score | 45 Days after the surgery
  impact of the robot assisted laparoscopy compared to conventional laparoscopy and by surgical laparotomy on the erectile function assessed by he EPIC 50 score (Expanded Prostate Cancer Index Composite)
impact of the robot assisted laparoscopy in prostatectomy on the urinary function assessed by EPIC 50 SCORE | up to 5 years after surgery
impact of the robot assisted laparoscopy in prostatectomy on the erectile function assessed by the International Index of Erectile Function (IIEF-5) score | upt to 5 years after the surgery
Assessment of the cost effectiveness of the robot assisted procedure in prostatectomy assessed by EQ5d-5L score | 12 months
  Assessment of the cost effectiveness of the robot assisted procedure in prostatectomy assessed by EQ5d-5L score
Occurence of prostatectomy sequelae (urinary incontinence or erectile dysfunction ) | 3 years
Occurence of prostatectomy sequelae (urinary incontinence or erectil dysfunction ) | 5 years
Prostate Specific Antigen (PSA) level | up to 5 years
  measures of the level of PSA in a man's blood

CONTACTS AND LOCATIONS:
Overall Officials: Shahnaz KLOUCHE, MD, Study Director — Elsan; Pierre-Thierry PIECHAUD, MD, Principal Investigator — Elsan
Locations (30):
- France (30):
  - Clinique Esquirol Saint Hilaire, Agen
  - Clinique Rhône Durance, Avignon
  - Hôpital Privé La Châtaigneraie, Beaumont
  - Clinique St Vincent, Besançon
  - Polyclinique de Franche Comté, Besançon
  - Clinique de Saint Augustin, Bordeaux
  - Clinique Keraudren - CHPB, Brest
  - Centre Médico-Chirurgical Les Cèdres, Brive-la-Gaillarde
  - Polyclinique Médipôle Saint-Roch, Cabestany
  - Polyclinique du Parc, Caen
  - Polyclinique Montréal, Carcassonne
  - Pôle Santé République, Clermont-Ferrand
  - Hôpital Privé Saint-François, Désertines
  - Clinique Cap-d'Or, La Seyne-sur-Mer
  - Pôle Santé Sud, Le Mans
  - Clinique Emailleurs-Colombier, Limoges
  - Polyclinique de Limoges, Limoges
  - Clinique Claude Bernard, Metz
  - Polyclinique de Gentilly, Nancy
  - Clinique Saint-Augustin, Nantes
  - Polyclinique Grand Sud, Nîmes
  - Polyclinique Les Fleurs, Ollioules
  - Polyclinique de Poitiers, Poitiers
  - Clinique du Renaison, Roanne
  - Clinique Guillaume De Varye, Saint-Doulchard
  - Centre clinical, Soyaux
  - Clinique de l'Estrée, Stains
  - Clinique Ambroise Paré, Toulouse
  - Polyclinique Vauban, Valenciennes
  - Hôpital privé Océane, Vannes

IPD SHARING:
Plan to Share IPD: Undecided